CLINICAL TRIAL: NCT00692952
Title: Effectiveness of BenZalkonium Chloride Gel as Vaginal Contraceptive: a Multicentric Randomized Controlled Trial
Acronym: BZK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Institute of Planned Parenthood Research (Other Government)
Collaborators: Shanghai Municipal Commission of Health and Family Planning (Other); Fudan University (Other); International Peace Maternity and Child Health Hospital (Other); Shanghai No. 1 Maternity and Child Care Center (Unknown); Chang Jiang Bio-pharmaceutical Co., Ltd. (Industry)
Responsible Party: Prof. Dr. Xuncheng DING, Shanghai Institute of Planned Parenthood Research
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: China FDA 2003L02778; ISRCTN16203579
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2009-07-10 (Estimated); Status verified 2008-06

CONDITIONS: Healthy
Keywords: contraceptive efficacy
MeSH Terms: interventions — Nonoxynol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 120 subjects using BenZalkonium Chloride Contraceptive Gel
  Interventions: Drug: a novel Benzalkonium Chloride (BZK) contraceptive gel
- 2 (Active Comparator): 120 subjects using Nonoxynol-9 contraceptive gel
  Interventions: Drug: LELEMI® contraceptive gel containing 50mg nonoxynol-9

INTERVENTIONS:
Drug: a novel Benzalkonium Chloride (BZK) contraceptive gel — insert 1 piece of the gel (containing 18mg BZK) into vagina before every coital act.
  Arms: 1
Drug: LELEMI® contraceptive gel containing 50mg nonoxynol-9 — insert 1 piece ofLELEMI® contraceptive gel within half an hour before every coital act
  Arms: 2

SUMMARY:
A multicentric clinical trial in three Chinese Maternal and Child Hospitals was conducted to evaluate the efficacy, safety and acceptability of newly-developed vaginal contraceptive gel, the optimized benzalkonium chloride (BZK) gel containing 18mg BZK, with comparison to a currently marketed (in China)contraceptive gel LELEMI® containing 50mg Nonoxynol-9 (N-9).

DETAILED DESCRIPTION:
A phase II, multicentric,randomized, controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* at risk for pregnancy and desiring contraception
* having regular menstrual cycle (21-35 days)
* at low risk for HIV or other sexually transmitted infection
* sexually active
* use the test products as their primary method of contraception
* keep a diary of coital activity, product use, and adverse events

Exclusion Criteria:

* diagnosis of any vaginal infection or any symptom of STDs at baseline
* known allergy or hypersensitivity to N-9 or BZK
* menopause for more than one month
* breastfeeding
* vaginal bleeding with unknown reasons
* genitourinary system anomaly
* hysteroptosis II or severe cystocele
* moderate to severe erosion of cervix
* malignant reproductive system tumors

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2004-03; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
contraceptive efficacy | March 2004 - November 2005

SECONDARY OUTCOMES:
acceptability | March 2004 - November 2005

CONTACTS AND LOCATIONS:
Overall Officials: Jinxun XU, MD, Principal Investigator — Shanghai Municipal Commission of Health and Family Planning
Locations (3):
- China (3):
  - Gynecology and Obstetrics Hospital of Fudan University, Shanghai
  - International Peace Maternity and Child Care Center, Shanghai
  - Shanghai No. 1 Maternity and Child Care Center, Shanghai